CLINICAL TRIAL: NCT02085096
Title: Problem-Solving Therapy for Prostate Cancer Patient's Spousal Caregivers
Brief Title: Problem Solving Therapy for Prostate Cancer Spousal Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: San Diego State University (Other)
Responsible Party: Principal Investigator, Georgia Robins Sadler, Professor, University of California, San Diego
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 5180
Record Dates: First submitted 2014-03-10; First posted 2014-03-12 (Estimated); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Prostate Cancer
Keywords: Caregivers; Coping Skills
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Problem-Solving Therapy (Experimental): A problem-solving therapy training program will be provided to the spouses/significant others of men diagnosed with prostate cancer. The purpose of this study is to test the efficacy of problem-solving therapy on the spouses of prostate cancer patients.
  Interventions: Behavioral: Problem-Solving Therapy
- Standard Supportive Care (Placebo Comparator): Participants who are randomized to this arm will be encouraged to use whatever supporting care is recommended to them by their health provider.
  Interventions: Behavioral: Problem-Solving Therapy

INTERVENTIONS:
Behavioral: Problem-Solving Therapy — Problem-solving therapy programs have been shown to be effective among parents of children diagnosed with cancer. Efforts have been made to apply this same strategy to spouses/significant others of men diagnosed with prostate cancer. The purpose of this study is to test the efficacy of problem-solving therapy on the spouses of prostate cancer patients.

SUMMARY:
Problem-solving therapy programs have been shown to be effective among parents of children diagnosed with cancer. Efforts have been made to apply this same strategy to spouses/significant others of men diagnosed with prostate cancer. The purpose of this study is to test the efficacy of problem-solving therapy on the spouses of prostate cancer patients.

DETAILED DESCRIPTION:
Problem-solving therapy programs have been shown to be effective among parents of children diagnosed with cancer. Efforts have been made to apply this same strategy to spouses/significant others of men diagnosed with prostate cancer. The purpose of this study is to test the efficacy of problem-solving therapy on the spouses of prostate cancer patients.

Participants were randomly assigned to an experimental group which received problem-solving therapy, or to a control group which relied on their standard methods of coping (e.g. their normal therapist, family and friends).

Participants completed baseline surveys regarding their distress and coping prior to randomization. They then completed these surveys again at post-intervention (approximately 2-3 months post-baseline) and 6 months post-baseline to determine lasting effects of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with prostate cancer within 18 months of study enrollment.
* The patient and significant other cohabited
* Couples resided in San Diego County
* Both patient and significant other were sufficiently proficient in English

Exclusion Criteria:

-

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 1997-07; Primary Completion 2002-12 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Change from Baseline of Effects of Stress and Coping to Follow-ups | From baseline to follow-ups at post-intervention (2-3 months post-baseline) and 6-months post-baseline

CONTACTS AND LOCATIONS:
Overall Officials: Georgia R Sadler, PhD, Principal Investigator — UC San Diego Moores Cancer Center; Vanessa L Malcarne, PhD, Principal Investigator — San Diego State University
Locations (1):
- UC San Diego Moores Cancer Center, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Banthia R, Malcarne VL, Varni JW, Ko CM, Sadler GR, Greenbergs HL. The effects of dyadic strength and coping styles on psychological distress in couples faced with prostate cancer. J Behav Med. 2003 Feb;26(1):31-52. doi: 10.1023/a:1021743005541. PMID 12690945
- [Background] Ko CM, Malcarne VL, Varni JW, Roesch SC, Banthia R, Greenbergs HL, Sadler GR. Problem-solving and distress in prostate cancer patients and their spousal caregivers. Support Care Cancer. 2005 Jun;13(6):367-74. doi: 10.1007/s00520-004-0748-5. Epub 2005 Jan 19. PMID 15657688
- [Background] Hawes S, Malcarne V, Ko C, Sadler G, Banthuia R, Sherman S, Varni J, Schmidt J. Identifying problems faced by spouses and partners of patients with prostate cancer. Oncol Nurs Forum. 2006 Jul 1;33(4):807-14. doi: 10.1188/06.ONF.807-814. PMID 16858462
- [Background] Yoshimoto SM, Ghorbani S, Baer JM, Cheng KW, Banthia R, Malcarne VL, Sadler GR, Ko CM, Greenbergs HL, Varni JW. Religious coping and problem-solving by couples faced with prostate cancer. Eur J Cancer Care (Engl). 2006 Dec;15(5):481-8. doi: 10.1111/j.1365-2354.2006.00700.x. PMID 17177907
- [Background] Merz EL, Malcarne VL, Ko CM, Sadler M, Kwack L, Varni JW, Sadler GR. Dyadic concordance among prostate cancer patients and their partners and health-related quality of life: does it matter? Psychol Health. 2011 Jun;26(6):651-66. doi: 10.1080/08870441003721251. Epub 2011 Jul 11. PMID 20680885